CLINICAL TRIAL: NCT00910195
Title: Validation of a New Automatic Bi-level Algorithm in the Treatment of Sleep-disordered Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Prof. Dr. Randerath, Institut für Pneumologie an der Universität Witten/Herdecke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: WI_BiLevel APAP_34/2008
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; CPAP; Bi-Level
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP before Bi-Level-APAP (Experimental): receiving CPAP treatment during the first night and then Bi-level-APAP treatment during second night
  Interventions: Device: CPAP treatment with subsequent Bi-Level-APAP treatment
- Bi-Level-APAP before CPAP (Experimental): receiving Bi-level-APAP treatment during the first night and then CPAP treatment during the second night
  Interventions: Device: Bi-Level-APAP treatment with subsequent CPAP treatment

INTERVENTIONS:
Device: CPAP treatment with subsequent Bi-Level-APAP treatment — CPAP treatment during the first night and then Bi-level-APAP treatment during second night
  Arms: CPAP before Bi-Level-APAP
Device: Bi-Level-APAP treatment with subsequent CPAP treatment — Bi-level-APAP treatment during the first night and then CPAP treatment during the second night
  Arms: Bi-Level-APAP before CPAP

SUMMARY:
Between 2%-4% of adult population suffers from obstructive sleep apnea (OSAS)(1), which is characterized by obstructive snoring, repetitive apnea and hypopnea in sleep, repetitive cyclic oxygen saturation, as a result from sleep fragmentation related to the arousals in sleeping profile and clinical consequences like day drowsiness, neuropsychological deficits, raised danger of accidents and cardiovascular disease. (1-6). The therapy of choice is the application of nasal continuous positive airway pressure (CPAP) (7-9).

Increasing relevance obtain the combined sleep-related breathing disturbances, where the patient shows an obstructive sleep apnea syndrome and some central breathing disturbances in the polysomnography at night. Those patients frequently present with cardiovascular diseases. These combined night breathing disturbances are frequently insufficient to be mitigated exclusively with a CPAP therapy.

Some modifications of nCPAP therapy were developed in order to optimize the therapy-compliance and the effectiveness of the therapy. Bi-level-CPAP-devices produce two pressure levels: one for inspiration and another for expiration, so that the patients are able expire against a constant low pressure. An increase in the use of this application in comparison between the conventional or the automatic CPAP therapy could not be proved in early studies. (12, 13) The principle of the automatic nCPAP therapy is to recognize the patient's current need of pressure and to alter the pressure within a set range by applying different algorithms. Some studies have shown that this therapy increased compliance and comfort (14-16), while other studies could not confirm these results. (17, 18)

The result of the current study should prove if the treatment of a new algorithm therapy based on an automatic bi-level-system for patients with sleep-related respiratory disorders is as effectively and subjective more comfortable as the conventional CPAP therapy.

Patients with a particularly high need of pressure should experience a clear expiratory pressure relief and a higher comfort. Therefore a better compliance is to expect. In the same way patients with additional central respiratory disturbances should obtain a benefit from the bi-level modus. This new treatment would help particularly such "critical patients", who are not responding well to the CPAP therapy or find it uncomfortable.

DETAILED DESCRIPTION:
Patients who meet all the above mentioned criteria and who were diagnosed as sleep-apnea syndrome patients in our hospital were asked to participate in the study. By a declaration of consent the patients were randomized in two different groups.

Group 1: started with CPAP at the first night and continued with Bi-level- APAP at the second night.

Group 2: began with Bi-level-APAP and ended with CPAP

Patients will be discharged with CPAP after the second night

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years.
* Newly diagnosed of sleep-apnea-syndrome, AHI> 5 per hour associated with the usual manifestation of this syndrome.
* Declaration of consent.

Exclusion Criteria:

* Absence of declaration of consent.
* Other relevant sleep disorders like insomnia, restless legs, parasomnia
* Heart failure NYHA-CLASS III- IV.
* Myocardial infarction or unstable angina pectoris or cardiac surgery in within the last three months.
* Apnea-hypopnea-index < 5 per hour.
* Pregnancy.
* Malign diseases.
* Serious chronic oxygen-requiring pulmonary illness.
* Age under 18 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Obstructive and central apnea-hypopnea-Index. | day one and two of the study

SECONDARY OUTCOMES:
Total apnea-hypopnea-index, minimum and middle oxygen saturation, subjective satisfaction with the therapy (questionnaire). | day one and two of the study

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Galetke, PD Dr., Study Chair; Winfried J. Randerath, Prof. Dr., Study Director
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, O'Connor GT, Boland LL, Schwartz JE, Samet JM. Sleep-disordered breathing and cardiovascular disease: cross-sectional results of the Sleep Heart Health Study. Am J Respir Crit Care Med. 2001 Jan;163(1):19-25. doi: 10.1164/ajrccm.163.1.2001008. PMID 11208620
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Finn L, Young T, Palta M, Fryback DG. Sleep-disordered breathing and self-reported general health status in the Wisconsin Sleep Cohort Study. Sleep. 1998 Nov 1;21(7):701-6. PMID 11286346
- [Background] Engleman HM, Kingshott RN, Martin SE, Douglas NJ. Cognitive function in the sleep apnea/hypopnea syndrome (SAHS). Sleep. 2000 Jun 15;23 Suppl 4:S102-8. PMID 10893080
- [Background] George CF. Sleep. 5: Driving and automobile crashes in patients with obstructive sleep apnoea/hypopnoea syndrome. Thorax. 2004 Sep;59(9):804-7. doi: 10.1136/thx.2003.007187. PMID 15333860
- [Background] Randerath WJ, Schraeder O, Galetke W, Feldmeyer F, Ruhle KH. Autoadjusting CPAP therapy based on impedance efficacy, compliance and acceptance. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):652-7. doi: 10.1164/ajrccm.163.3.2006168. PMID 11254519
- [Background] Randerath WJ, Galetke W, Ruhle KH. Auto-adjusting CPAP based on impedance versus bilevel pressure in difficult-to-treat sleep apnea syndrome: a prospective randomized crossover study. Med Sci Monit. 2003 Aug;9(8):CR353-8. PMID 12942031